CLINICAL TRIAL: NCT03817684
Title: A Randomized , Double Blind, Placebo Controlled, 3-Arm Parallel Design Study to Evaluate the Effects of BPN14770 in Patients With Early Stage Alzheimer's Disease
Brief Title: Tetra PICASSO AD Trial: Study to Evaluate Effects of BPN14770 in Early Alzheimer's Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPN14770-CNS-201
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BPN14770 10mg bid (Experimental): 10 mg bid dose of the Drug BPN14770
  Interventions: Drug: BPN14770
- BPN 14770 25mg bid (Experimental): 25mg bid dose of the Drug BPN14770
  Interventions: Drug: BPN14770
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPN14770 — Drug BPN14770
  Arms: BPN 14770 25mg bid; BPN14770 10mg bid
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo Controlled, 3-Arm Parallel Design Study to Evaluate the Effects of BPN14770 in Patients with Early Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 55 and 85 years with a clinical diagnosis of early stage AD, defined according to the following criteria assessed during Screening and at Baseline :

   1. Clinical Dementia Rating (CDR) score of 0.5 or 1, with Memory Box score of 0.5 or greater
   2. MMSE score of 20 or greater
   3. RBANS DMI score ≤ 85 Note: PET imaging for amyloid is not required for diagnosis, which will be made on clinical grounds.
2. Currently receiving a stable (at least 2 months) dose regimen of donepezil or another cholinesterase inhibitor for treatment of Alzheimer's disease. Doses of these drugs may not be changed during the trial.

   Note: Memantine is not permitted during the trial and must be discontinued at least 3 weeks prior to Baseline.
3. Modified Hachinski Ischemia score < 4.
4. Body mass index (BMI) < 38 kg/m2, inclusive, and body weight of >48 kg (105 pounds) at screening.
5. Female subjects must be at least two years post-menopausal (subjected reported menopausal status), surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to first study drug administration), or willing to either (1) utilize hormonal contraception plus one barrier method or (2) use two barrier methods of contraception (e.g. diaphragm and spermicide) from initial screening until one month after taking the final dose. An intrauterine device (IUD) is considered a barrier method of contraception in this study. Male subjects must be willing to inform female partners of their participation in the study and must agree to use adequate contraceptive methods (vasectomy performed at least 6 months prior to first study drug administration, or use at least one barrier method of birth control).
6. Able to understand and comply with the study procedures, voluntarily agree to participate in this study, and provide written informed consent prior to start of any study-specific procedures.
7. All subjects must have a caregiver who is willing and able to ensure compliance with study medications, visits, and study procedures.

Exclusion Criteria:

1. Any medical or neurological condition (other than early stage AD) that might be a contributing cause to the subject's cognitive impairment.
2. History of stroke or multiple (>3 discreet episodes) Transient Ischemic Attacks (TIAs), severe head trauma with cognitive sequelae, uncontrolled seizures, or unexplained prolonged loss of consciousness (> 1 minute) during the past year.
3. Clinically significant major psychiatric illness during the past 6 months.
4. History of unstable angina, myocardial infarction, chronic heart failure, or clinically significant conduction abnormalities during the past year.
5. Clinically significant liver or renal disease.
6. Clinically significant abnormality, in the Investigator's judgment, in hematology, chemistry, or urinalysis.
7. Positive serology results for hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV).
8. Abnormal liver function test at the Screening Visit (aspartate aminotransferase or alanine aminotransferase >2

   × the upper limit of normal [ULN], or total bilirubin >1.7 × ULN, based on appropriate age and gender normal values). Subjects may be re-screened once.
9. Marked hypotension (systolic blood pressure [BP] ˂90 mmHg or diastolic BP ˂50 mmHg) or hypertension (systolic BP ˃160 mmHg or diastolic BP ˃100 mmHg) based on sitting values. O ut-of-range results may be repeated once at Screening, and eligibility must be confirmed at Baseline.
10. Marked bradycardia (heart rate ˂45 beats per minute [bpm]) or tachycardia (heart rate ˃115 bpm) based on supine ECG values. Out-of-range results may be repeated once at Screening, and eligibility must be confirmed at Baseline.
11. Clinically important conduction abnormalities on ECG, or evidence or history of long QT syndrome based on supine ECG values obtained at Screening. Out-of-range results may be repeated once and eligibility confirmed at Baseline.
12. Active gastric or duodenal ulcers or other diseases of the gastrointestinal tract that could interfere with absorption of study drug. Note: Subjects with a history of appendectomy or cholecystectomy may be enrolled.
13. Active acute or chronic infectious diseases that would interfere with subject's participation in the study.
14. Unable to discontinue centrally active medications (other than cholinesterase inhibitors), including memantine, psychotropic drugs other than SSRIs (which must have been stable for 2 months and remain stable throughout the study), sedative antihistamines or other centrally active medications with potential cognitive effects (e.g., CNS-penetrant beta blockers).
15. Unable to discontinue moderate to strong inhibitors or inducers of CYP3A4, CYP2D6, or other cytochromes at least 14 days prior to the first dose of study drug. A complete listing of such inhibitors or inducers may be found in http://medicine.iupui.edu/clinpharm/ddis/main-table (Other prescription or non-prescription drugs such as antihypertensive or cholesterol lowering agents are allowed, if, in the Investigator's judgement, they would not interfere with the study medication or the cognitive testing.)
16. A suicidal ideation intensity score of 3 or higher per screening Columbia Suicide Severity Rating Scale (CSSRS) assessment on Day 1 (Baseline) and/or any suicidal behavior within the past 28 days.
17. History of chronic alcohol or other substance abuse, including marijuana, within the previous year prior to the Screening visit (per the current edition of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5), or regular (daily) consumption of alcohol exceeding two bottles of beer, or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
18. Inability or unwillingness to comply with the protocol, including performing the cognitive function tests, or likely inability to complete the study.
19. Participation in other clinical studies involving investigational drug within the previous 30 days prior to the Screening Visit.
20. Donation of blood within 4 weeks, or blood products within 2 weeks, prior to first study drug administration.
21. History of clinically significant drug allergy that includes symptoms such as shortness of breath, rash, or edema.
22. Clinically significant B12 deficiency within 12 months prior to Visit 1 (Screening). Participants on stable replacement therapy for a minimum of 3 consecutive months immediately prior to Visit 1 (Screening) may be included

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reines, MD, Study Director — Tetra Discovery Partners
Locations (41):
- United States (41):
  - Generations at Agritopia/CCT Research, Gilbert, Arizona
  - CiTrials, Inc., Bellflower, California
  - ATP Clinical Research, Inc, Costa Mesa, California
  - Alliance for Research, Long Beach, California
  - Pacific Research Network Inc., San Diego, California
  - HB Clinical Trials, Inc., Santa Ana, California
  - Mile High Research Center, Denver, Colorado
  - JEM Research Insitute, Atlantis, Florida
  - Linfritz Research Group, Coral Gables, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Galiz Research, Hialeah, Florida
  - Alzheimer's Research and Treatement Center, Lake Worth, Florida
  - Optimus Clinical Research, Miami, Florida
  - BioMed Research Institute, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - Arocha Research Center, Miami, Florida
  - Allied Biomedical Research Institute Inc., Miami, Florida
  - Advanced Clinical Research Network, Miami, Florida
  - Gutierrez Medical Center LLD, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Palm Beach Neurological Center, Palm Beach, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Synergy Clinical Research, Pensacola, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Neurosciences Research, Elk Grove Village, Illinois
  - Hassman Research Institute, Berlin, New Jersey
  - Advanced Memory Research Institute of NJ PC, Toms River, New Jersey
  - Integrative Clinical Trials, Brooklyn, New York
  - Neurological Associates of Long Island, Lake Success, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - Alzheimers Memory Center, Charlotte, North Carolina
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - MDH Research, Westerville, Ohio
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Aspen Clinical Research, Orem, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BPN14770 10mg Bid: 10 mg bid dose of the Drug BPN14770 BPN14770: Drug BPN14770
- BPN 14770 25mg Bid: 25mg bid dose of the Drug BPN14770 BPN14770: Drug BPN14770
Period: Overall Study
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Started | 84 | 85 | 86
Safety Population (All randomized participants who received at least 1 dose of study treatment.) | 80 | 85 | 86
Completed | 79 | 79 | 84
Not Completed | 5 | 6 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo | Total
Number analyzed (Participants) | 80 | 85 | 86 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (7.54) | 71.8 (7.21) | 71.2 (7.65) | 71.3 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 58 | 51 | 154
  Male | 35 | 27 | 35 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 54 | 50 | 148
  Not Hispanic or Latino | 36 | 31 | 36 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 9 | 25
  White | 70 | 78 | 77 | 225
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 85 | 86 | 251
Pre Treatment MMSE [Mean (Standard Deviation); unit: scores on a scale] — The MMSE consisted of 11 items covering orientation, memory (recent and immediate), concentration, language and praxis. Total score ranges from 0 (severe cognitive impairment) to 30 (intact cognitive function), with lower scores indicating greater cognitive impairment. In participants with a diagnosis of Alzheimer's Disease (AD), lower scores indicating worse disease. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
  scores on a scale | 24.2 (2.04) | 24.3 (2.61) | 24.6 (2.44) | 24.4 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neurological Status- Delayed Memory Index (RBANS- DMI) at Week 13
Description: The RBANS is a brief, individually administered test measuring attention, language, visuospatial/constructional abilities, and immediate and delayed memory. It consists of 12 subtests, which yield 5 Index scores and a Total Scale score. Lower scores indicate worse performance on the test (and thus greater impairment). Scores for the RBANS DMI range from 40 (greater impairment) to 160 (improved function), with higher scores indicating improved function.
Time Frame: Baseline, Week 13
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 10.1 (1.71) | 9.9 (1.67) | 9.7 (1.63)

2. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neurological Status (RBANS) Total Score at Week 13
Description: The RBANS is a brief, individually administered test measuring attention, language, visuospatial/constructional abilities, and immediate and delayed memory. It consists of 12 subtests, which yield 5 Index scores and a Total Scale score. Lower scores indicate worse performance on the test (and thus greater impairment). The RBANS total score ranges from 40 to 160, with higher scores indicating improved function.
Time Frame: Baseline, Week 13
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 4.5 (0.98) | 5.2 (0.96) | 5.4 (0.94)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) Total Score at Week 13
Description: The ADCS-ADL is an interviewer-administered informant-based scale where the informant (caregiver) responds to 23 activities of daily living questions about the participant. The questions range from basic to instrumental activities of daily living. The total score ranges from 0-78 and a higher score signifies greater functional ability.
Time Frame: Baseline, Week 13
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 1.1 (0.55) | 1.5 (0.54) | 1.5 (0.53)

4. Secondary Outcome: Change From Baseline in Mini-Mental State Exam (MMSE) Total Score at Week 13
Description: The MMSE consists of 11 items covering orientation, memory (recent and immediate), concentration, language and praxis. Total score ranges from 0 (severe cognitive impairment) to 30 (intact cognitive function), with lower scores indicating greater cognitive impairment. In participants with a diagnosis of AD, lower scores indicating worse disease. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
Time Frame: Baseline, Week 13
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 0.7 (0.23) | 0.8 (0.23) | 0.8 (0.23)

5. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes Score (CDR-SB) at Week 13
Description: The CDR was developed primarily to assess severity level in persons with dementia. Six domains were assessed and then synthesized to assign a Global CDR score. The domains were memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Impairment was defined only when caused by cognitive loss rather than by physical disability or other non-cognitive factors. CDR is an ordinal parameter (scale 0 [least impairment]-3 [severe impairment]). CDR-SB score was obtained by summing each of the domain box scores, with scores ranging from 0 (least impairment) to 18 (severe impairment).
Time Frame: Baseline, Week 13
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 0.25 (0.119) | -0.05 (0.118) | 0.19 (0.114)

6. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The Investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse.
Time Frame: Week 13
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
Number analyzed (Participants) | 80 | 84 | 86
scores on a scale | 3.5 (0.10) | 3.3 (0.10) | 3.4 (0.10)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | BPN14770 10mg Bid | BPN 14770 25mg Bid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/85 | 0/86
Serious Adverse Events (participants affected / at risk) | 2/80 | 2/85 | 2/86
Other Adverse Events (participants affected / at risk) | 9/80 | 11/85 | 3/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPN14770 10mg Bid (N=80) | BPN 14770 25mg Bid (N=85) | Placebo (N=86)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolsis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral Neck Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPN14770 10mg Bid (N=80) | BPN 14770 25mg Bid (N=85) | Placebo (N=86)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03817684/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03817684/SAP_003.pdf